CLINICAL TRIAL: NCT02427282
Title: Miniscrew-supported Versus Standard Frog Molar Distalizing Appliances (Clinical Study)
Brief Title: Distalization by Miniscrew
Acronym: AU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Riyadh Abdullah Iskander, PhD candidate, orthodontic department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 999
Record Dates: First submitted 2015-04-19; First posted 2015-04-28 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Distalization by Miniscrews

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MS. Frog (Active Comparator): miniscrew-supported frog molar distalizing appliance
  Interventions: Device: miniscrew-supported Frog molar distalizing appliance
- Stand. Frog (Experimental): Standard Frog appliance
  Interventions: Device: Standard Frog molar distalizing appliance

INTERVENTIONS:
Device: miniscrew-supported Frog molar distalizing appliance — miniscrew 10mm length and 1.7mm diameter FORESTADENT company
  Other Names: Skeletal Frog
  Arms: MS. Frog
Device: Standard Frog molar distalizing appliance — Nance buttons attached to first premolars band
  Other Names: Conventional Frog
  Arms: Stand. Frog

SUMMARY:
This study aimed to compare the effectiveness and efficiency of miniscrew-supported and standard frog molar distalizing appliances.

DETAILED DESCRIPTION:
A prospective randomized clinical trial study was carried out on twenty healthy Egyptian subjects, each required molar distalization as part of their comprehensive orthodontic treatment. The subjects were selected and treated at the outpatient clinic of the Orthodontic Department, Faculty of Dentistry, Ain-Shams University.

The inclusion criteria in this subject selection in this study was as follows;

1. All the subjects had an age range from 11 to 16 years with a mean of ±13.5 years.
2. All the subjects had skeletal Class 1 or mild skeletal Class 2 due to maxillary excess.
3. All the subjects had bilateral Class II molar relationship.
4. All subjects were free from any dental anomalies.
5. All subjects had good oral hygiene. The exclusion criteria in this study was as follows; 1- Missing permanent teeth with exception of 3rd molar. 2- Previous orthodontic treatment. 3- Systemic disease that may influence orthodontic treatment and drug intake. 4- Periodontal disease. 5- Functional mandibular deviations and facial asymmetry. 6- History of parafunctional habits.

The subjects were equally and randomly divided into two groups; group A and group B which included ten subjects per group. These groups were classified according to the type of distalizer utilized:

* Group A: included ten subjects utilizing the conventional frog molar distalizing appliance (CF).
* Group B: included ten subjects utilizing the Miniscrews-supported frog molar distalizing appliance (MSF)

The pretreatment and post-distalization Database Records All subjects had the following records; a clinical diagnostic sheet, orthodontic study cast (according to ABO index), extraoral and intraoral photographs, and CBCT.

These records were obtained at T1 before distalization and at T2 after distalization.

The study protocol was approved by the local ethics committee, faculty of dentistry, Ain-Shams University. Before commencing with treatment, all the subjects and their guardians received a full explanation of the treatment protocol. After which they were asked to sign a detailed written consent.

ELIGIBILITY:
Inclusion Criteria:

1. All the subjects had an age range from 11 to 16 years with a mean of ±13.5 years.
2. All the subjects had skeletal Class 1 or mild skeletal Class 2 due to maxillary excess.
3. All the subjects had bilateral Class II molar relationship.
4. All subjects were free from any dental anomalies.
5. All subjects had good oral hygiene.

Exclusion Criteria:

1. Missing permanent teeth with exception of 3rd molar.
2. Previous orthodontic treatment.
3. Systemic disease that may influence orthodontic treatment and drug intake.
4. Periodontal disease.
5. Functional mandibular deviations and facial asymmetry.
6. History of parafunctional habits.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
mesial migration of anterior teeth measured in millimeter and angles by using cone beam computerized tomography | 6months
  pretreatment and postdistalization records as cone beam computerized tomography and cast analysis